CLINICAL TRIAL: NCT01486797
Title: A Multi-center, Open Label, Uncontrolled, Phase IIA Clinical Trial Evaluating the Safety and Efficacy of NOX A12 in Combination With a Background Therapy of Bendamustine and Rituximab (BR) in Previously Treated Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: NOX-A12 in Combination With Bendamustine and Rituximab in Relapsed Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNOXA12C201; 2011-004672-11 (EudraCT Number)
Record Dates: First submitted 2011-12-01; First posted 2011-12-07 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Relapsed Chronic Lymphocytic Leukemia (CLL); NOX-A12; Bendamustine; Rituximab; Spiegelmer; Chemosensitization; Stromal cell-derived factor-1 (SDF-1); CXCL12
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — NOX-A12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NOX-A12 (Experimental)
  Interventions: Drug: NOX-A12

INTERVENTIONS:
Drug: NOX-A12 — Pilot Group (NOX-A12 single agent, and combined with BR):
  * 3 cohorts of 3 patients will receive treatment with NOX-A12 alone at a single dose of 1, 2 or 4 mg/kg i.v. 2 weeks before the combination treatment of NOX-A12 and BR begins.The combination of NOX-A12 and BR will follow a dose titration design beginning at 1 mg/kg NOX-A12 (cycle 1), proceeding to dose levels of 2 mg/kg (cycle 2) and 4 mg/kg (cycle 3) NOX-A12 in combination with BR. This is followed by consolidation in cycles 4-6 when NOX-A12 will be kept at the highest individually titrated dose.
  Expansion Group (NOX-A12 in combination with BR):
  * Expansion patients will not receive single agent NOX-A12, but will receive combination treatment as for the pilot group.
  Other Names: olaptesed pegol

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of NOX A12 in combination with a background therapy of bendamustine and rituximab (BR) chemotherapy in previously treated patients with chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
CLL cells express high levels of CXCR4 chemokine receptors, which cause leukemia cell migration and adhesion to stromal cells secreting the CXCR4 ligand, CXCL12 (or stromal-derived-factor 1, SDF-1). NOX A12 is a specific CXCL12 antagonist and may improve BR therapy by disrupting CXCR4-CXCL12 interactions, thereby mobilizing CLL cells from protective tissue microenvironments to the blood. Furthermore, SDF-1 inhibition may alter the activation status of CLL cells, thereby triggering apoptosis or sensitization of CLL cells towards chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of B-cell CLL
2. Relapsed, bendamustine-sensitive (at least partial response with a duration of at least six months) or bendamustine-naive patients after at least one but not more than 3 prior treatments of their disease.
3. CLL in need of treatment (Binet C or A/B with active disease) according to Hallek et al. 2008
4. Subject must have measurable disease according to NCI-WG criteria (for details see Hallek M, Blood 2008; 111: 5446-5456).
5. Pre-study WHO performance status ≤ 2 and modified cumulative illness rating score (CIRS) of less than 7.
6. Signed, written informed consent.
7. Men and women of reproductive potential must agree to follow accepted birth control methods during treatment and for 3 months after completion of treatment.
8. Acceptable liver function: Bilirubin ≤ 1.5 x upper limit of normal (ULN) at screening, AST (SGOT) and/or ALT (SGPT) ≤ 2.5 x ULN.
9. Acceptable hematologic status: Platelet count ≥ 75 x 109/L, ANC > 0.75x109/L.
10. Acceptable renal function: Serum creatinine ≤1.5 ULN and/or calculated creatinine clearance (Cockroft-Gault Formula) ≥ 50 mL/min
11. Male or female, age ≥ 18
12. No clinically significant abnormalities of liver volume, liver hemodynamics or elasticity, measured by abdominal ultrasound.

Exclusion Criteria:

1. Relapse of B-cell CLL within 12 months after last chemotherapy.
2. Subjects who have progressed to more aggressive B-cell cancers such as Richter's syndrome.
3. CLL with documented loss of the short arm of chromosome 17 (17p-) associated with the loss of p53.
4. The subject has a history of or is clinically suspicious for cancer-related Central Nervous System disease.
5. Patients at risk of hemostasis or spleen rupture.
6. Autoimmune hemolytic anemia.
7. Prior allogeneic stem cell transplant (alloSCT) or patients who are considered to be candidates for allo SCT as assessed by their treating physician
8. Patient has a history of other active malignancies within three years prior to study entry, with the exception of: adequately treated in situ carcinoma of the cervix uteri; basal or squamous cell carcinoma of the skin; in situ carcinoma of the bladder; previous malignancy confined and surgically resected with curative intent.
9. The patient exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to: uncontrolled systemic infection (viral, bacterial, or fungal); diagnosis of fever and neutropenia within 1 week prior to study drug administration.
10. Female subject is pregnant or breast-feeding.
11. Known infection with HIV, active Hepatitis B or Hepatitis C.
12. The patient has a history of prior toxicity from bendamustine or rituximab that resulted in permanent discontinuation of treatments.
13. Treatment with other investigational drugs, or participation in another clinical trial within 30 days prior to study drug administration.
14. Uncontrolled hypertension (defined as systolic blood pressure (BP) > 160 mm Hg or diastolic BP > 100 mm Hg).
15. Myocardial infarction or unstable angina within the past 6 months prior to study drug administration.
16. Systemic illnesses or other severe concurrent disease including alcoholism which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and efficacy of the investigational treatments.
17. Known or suspected of not being able to comply with the trial protocol.
18. Having been previously enrolled in this clinical trial.
19. Known hypersensitivity to rituximab or to any of the excipients or to murine proteins
20. History of recurring or chronic infections or underlying conditions which may further predispose patients to serious infection.
21. Known hypersensitivity to bendamustine or to mannitol.
22. Invasive surgery within 30 days prior to study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of NOX A12 alone and in combination with BR. | 30 months
  The safety evaluation will be based on the following assessments:
  * adverse events
  * vital signs
  * 12 lead ECGs
  * laboratory parameters
  * immunogenicity
Complete remission (CR) rate | 6 months
  Assessment of the complete remission rate after cycle 3 and 6 will be the primary efficacy endpoint. The 1996 NCI-WG criteria which have been updated in 2008 will be applied.

SECONDARY OUTCOMES:
Pharmacodynamics of NOX-A12 alone and in combination with BR | 6 months
  The pharmacodynamics evaluation will be based on the following assessments:
  * mobilization of peripheral blood CD34+ cells and CLL cells
  * plasma concentration of SDF-1/CXCL12
Overall response rate (ORR = CR + PR) | 6 months
Progression free survival (PFS) | 30 months
Pharmacokinetics of NOX-A12 alone and in combination with BR | 10 time points over 6 months
  The pharmacokinetics evaluation will be based on the following assessments:
  * plasma concentration of NOX-A12
  * 24-hour urine excretion of NOX-A12
Event free survival (EFS) | 30 months
Time to progression (TTP) | 30 months
Duration of response (DOR) | 30 months
Overall survival (OS) | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Kai Riecke, MD, Study Director — TME Pharma AG
Locations (17):
- Austria (4):
  - Medical University Innsbruck, Division of Hematology and Oncology, Innsbruck
  - University Hospital Salzburg, Department of Medicine III, Center of Oncology and Hematology, Salzburg
  - Landeskrankenhaus Steyr, Department of Internal Medicine II (Hematology and Oncology), Steyr
  - Hospital Wels-Grieskrichen, Department of Internal Medicine IV (Hematology and Oncology), Wels
- Belgium (3):
  - Cliniques universitaires Saint-Luc, Brussels
  - Institute Jules Bordet, Department of Hematology, Brussels
  - University Hospital Gasthuisberg, Department of Hematology, Leuven
- France (3):
  - Centre Hospitalier Universitaire Clémenceau, Department of Hematology, Caen
  - Hospices Civils, Department of Hematology, Lyon
  - Centre Hospitalier Universitaire de la Milétrie, Department of Hematology, Poitiers
- Italy (7):
  - University Hospital, Institute of Hematology and Oncology, Bologna
  - Azienda Sanitaria Locale 8, Department of Oncology, Cagliari
  - University Hospital San Martino, Department of Hematology and Oncology, Genova
  - Niguarda Ca'Granda Hospital, Milan
  - University Scientific Research Institute San Raffaele, Milan
  - University School of Medicine, Department of Hematology, Padua
  - University La Sapienza, Department of Cellular Biotechnologies and Hematology, Rome

REFERENCES:
- [Derived] Steurer M, Montillo M, Scarfo L, Mauro FR, Andel J, Wildner S, Trentin L, Janssens A, Burgstaller S, Fromming A, Dummler T, Riecke K, Baumann M, Beyer D, Vauleon S, Ghia P, Foa R, Caligaris-Cappio F, Gobbi M. Olaptesed pegol (NOX-A12) with bendamustine and rituximab: a phase IIa study in patients with relapsed/refractory chronic lymphocytic leukemia. Haematologica. 2019 Oct;104(10):2053-2060. doi: 10.3324/haematol.2018.205930. Epub 2019 May 16. PMID 31097627
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581